CLINICAL TRIAL: NCT01489709
Title: Specified Drug Use Results Survey of Vesicare Tablets
Brief Title: Post Marketing Survey of Vesicare in Japan
Acronym: SET-Q
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 905-JC-VC0004
Record Dates: First submitted 2011-12-08; First posted 2011-12-12 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Overactive Bladder
Keywords: overactive bladder; solifenacin; Overactive bladder questionnaire; Overactive Bladder Symptom Score; satisfaction score
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Vesicare group: Who receive vesicare
  Interventions: Drug: Vesicare

INTERVENTIONS:
Drug: Vesicare — oral
  Other Names: solifenacin

SUMMARY:
This study is to evaluate the effect of Vesicare on quality of life (QOL) in female patients.

DETAILED DESCRIPTION:
Overactive bladder (OAB) represents a constellation of symptoms that must include urinary urgency as an essential symptom for the diagnosis. It is usually accompanied by daytime frequency and nighttime frequency (urgency incontinence is not an essential symptom) and impairs the patient's activities of daily living and quality of life (QOL).

The objective of this survey is to confirm QOL improvement in patients treated with Vesicare (Generic Name: solifenacin succinate), with the use of OAB-q (Overactive bladder questionnaire), a questionnaire for assessment of OAB symptoms and QOL. The effect of improvement of OAB symptoms by solifenacin on QOL will also be confirmed. This survey will not include male OAB patients since many of them have benign prostatic hyperplasia as a coexisting disease and their QOL is supposed to be affected by α1-blocker treatment. To define patient's response to solifenacin in terms of QOL more clearly, this survey will include only female OAB patients.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated OAB patients
* Patients who meet the diagnostic criteria for OAB provided in the clinical guidelines for overactive bladder (patients who have urinary urgency at least once weekly as an essential symptom and at least one of the other OAB symptoms including daytime frequency, nighttime frequency, and urgency incontinence)
* Patients who can understand and answer OAB-q (Japanese version)
* Patients from whom data on all items concerning OABSS, OAB-q, and satisfaction score for urination can be obtained at baseline
* Patients who are expected to be treated for at least 12 weeks

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who meet the diagnostic criteria for OAB provided in the clinical guidelines for overactive bladder (patients who have urinary urgency at least once weekly as an essential symptom and at least one of the other OAB symptoms including daytime frequency, nighttime frequency, and urgency incontinence)
Sampling Method: Non-Probability Sample
Enrollment: 1160 (Actual)
Dates: Start 2010-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Changes in OAB-q (overactive bladder questionnaire) | Baseline and at 12 weeks (or last observation period)

SECONDARY OUTCOMES:
Changes in OABSS (overactive bladder symptom score) | Baseline and at 12 weeks (or last observation period)
Changes in satisfaction score for urination | Baseline and at 12 weeks (or last observation period)

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (8):
- Japan (8):
  - Chugoku
  - Chūbu
  - Hokkaido
  - Kansai
  - Kantou
  - Kyushu
  - Shikoku
  - Tōhoku